CLINICAL TRIAL: NCT05319444
Title: Cleansing Device for the Treatment of Scalp and Hair Conditions
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: This study has a patent application submitted to the patent office
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DERM-2021-29445
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Dandruff; Seborrheic Dermatitis; Hair Loss
MeSH Terms: conditions — Dandruff; Dermatitis, Seborrheic; Alopecia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (8):
- Healthy Scalp and one treatment (Experimental): Participants with healthy scalps who will receive one treatment with the device and complete one in-person follow-up.
  Interventions: Device: Off-brand Waterpik®
- Healthy Scalp and three treatments (Experimental): Participants with healthy scalps who will receive three treatments with the device and complete one in-person follow-up.
  Interventions: Device: Off-brand Waterpik®
- Dandruff and one treatment (Experimental): Participants with dandruff who will receive one treatment with the device and complete one in-person follow-up.
  Interventions: Device: Off-brand Waterpik®
- Dandruff and three treatments (Experimental): Participants with dandruff who will receive three treatments with the device and complete one in-person follow-up.
  Interventions: Device: Off-brand Waterpik®
- Hair loss disease and one treatment (Experimental): Participants with hair loss disease who will receive one treatment with the device and complete one in-person follow-up.
  Interventions: Device: Off-brand Waterpik®
- Seborrheic Dermatitis with one treatment (Experimental): Participants with seborrheic dermatitis disease who will receive one treatment with the device and complete one in-person follow-up.
  Interventions: Device: Off-brand Waterpik®
- Seborrheic Dermatitis and three treatments (Experimental): Participants with seborrheic dermatitis who will receive three treatments with the device and complete one in-person follow-up.
  Interventions: Device: Off-brand Waterpik®
- Hair loss disease and three treatments (Experimental): Participants with hair loss disease who will receive three treatments with the device and complete one in-person follow-up.
  Interventions: Device: Off-brand Waterpik®

INTERVENTIONS:
Device: Off-brand Waterpik® — Study staff will use the Waterpik® device and brush for approximately two to five minutes on the participant's scalp until all scale and other debris appears to be resolved. Their scalp will then be rinsed and gently dried with a towel.
  The off-label design utilizes the Waterpik® device, but with adjustments optimized for scalp health. The device settings are adjustable during the treatment, ranging from settings of 2-10. Study staff plan to utilize the setting of 10 unless the participant indicates discomfort. Investigators attached a small Losophy brush in replacement of the Waterpik® toothbrush. The small Losophy brush was connected to the device via PVC heat shrink and a hole was drilled on the brush in order to deliver water while simultaneously utilizing the brush on the scalp.

SUMMARY:
The objective of this study is to evaluate an improvement of scalp health after the use of an investigational off-label WaterPik and brush device aimed to massage and cleanse the scalp.

DETAILED DESCRIPTION:
Seborrheic dermatitis and dandruff are skin conditions that present with common features and respond similarly to treatments. Dandruff involves flaking skin that can cause irritation and itching. Dandruff only involves the scalp, whereas seborrheic dermatitis can occur on the scalp, face, chest, and retro-auricular areas. Seborrheic dermatitis can also result in itching and flaking, as well as inflammation and erythema. Both dandruff and seborrheic dermatitis are known to be harmful to the scalp.

Despite shampoo and washing, one may still continue to have flaking and scale present on the scalp. There are numerous scalp massages and brushes on the consumer market. Waterpik® was FDA approved in 2018 to provide pressured water combined with a powered toothbrush for optimal plaque and particle removal when cleaning the mouth and teeth. Waterpik® now has several products on the market designed for oral health, pet care, and washing in the shower. The off-label design utilizes the Waterpik® device, but with adjustments optimized for scalp health.

Through the investigational use of the off-label WaterPik® and brush device, the investigators propose the technique of massage and gentle water pressure will reduce seborrheic dermatitis and dandruff on the scalp.

ELIGIBILITY:
Inclusion Criteria:

* Participants must qualify for one of the following scalp conditions based on clinical opinion of a board-certified dermatologist: healthy scalp, dandruff, seborrheic dermatitis, or hair loss disease
* All Women of Child Bearing Potential must indicate use of two of the following contraceptive methods. The WaterPik device uses an ultrasonic technology which includes ultrasound. Unnecessary ultrasound is not recommended for pregnant women.

  * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal)
  * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable)
  * Intrauterine device (IUD)
  * Intraurerine hormone-releasing system (IUS)
  * Vasectomized partner
  * Sexual abstinence
  * Barrier method, such as a condom

Exclusion Criteria:

* Non-English speaking
* Exclusion related to pregnancy, lactation, or plans to become pregnant over the course of the study (based on self-report from the participant)
* Current clinical condition that, in the opinion of the site investigator, would interfere with adherence to study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in Adherent Scalp Flaking Scale (ASFS) | 4 weeks
  The presence of dandruff flakes adhereing to the scalp in 8 defined areas is rated on a scale of 0-10 per area, where 0 indicates no flakes and 10 indicates heavy flaking. This is combined for total scores ranging from 0-80.

SECONDARY OUTCOMES:
Change in Erythema Score | 4 weeks
  The presence of erythema is rated on a scale of 0-4, where 0 indicates None, 1 indicates Minimal - barely perceptible erythema, 2 indicates Mild - predominantly minimal erythema (pink) in the treated area with or without a few isolated areas of more intense erythema, 3 indicates Moderate - predominantly moderate erythema (red) in the treated area with or without a few isolated areas of intense erythema (bright red), and 4 indicates Severe - predominantly intense erythema (bright red) in the treated area with or without a few isolated areas of very intense (fiery red) erythema. The higher score means a worse outcome.
Change in Patient Sensory Assessment of Scalp & Hair Score | 4 weeks
  This Score is based on 12 descriptions that patients rate 0-10 to assess the condition of their scalp and hair. A higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ronda Farah, MD, Principal Investigator — University of Minnesota Medical School Department of Dermatology; Maria Hordinsky, MD, Principal Investigator — University of Minnesota Medical School Department of Dermatology
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No